CLINICAL TRIAL: NCT00783822
Title: Behavioral and Psychosocial Effects of Rapid Genetic Counseling and Testing in Newly Diagnosed Breast Cancer Patients: a Multicenter Study
Brief Title: Effects of Rapid Genetic Counseling and Testing in Newly Diagnosed Breast Cancer Patients
Acronym: TIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: UMC Utrecht (Other); Fonds NutsOhra (Other)
Responsible Party: Principal Investigator, Neil Aaronson, Head, Department of Psychosocial Research, Division of Psychosocial Research & Epidemiology, The Netherlands Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NL24252.031.08; SNO-T-0701-95
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Breast Neoplasms
Keywords: breast neoplasms; genetic counseling
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Other): rapid genetic counseling and testing
  Interventions: Other: RGCT
- control (No Intervention): usual care

INTERVENTIONS:
Other: RGCT — rapid genetic counseling and testing
  Arms: intervention

SUMMARY:
5-10% of breast cancer patients carry a mutation in the BRCA1 or BRCA2 gene. Genetic counseling and DNA testing are usually offered to selected patients after primary treatment has been completed (e.g. the first year after diagnosis). For women with a mutation in one of the two breast-ovarian cancer syndrome genes, chances of a second breast cancer are high, and therefore a proportion of these women may opt for preventive measures in addition to their immediate breast cancer treatment. Contralateral prophylactic mastectomy significantly reduces this risk, and is associated with a reduction in mortality.

Genetic counseling and testing for breast cancer typically takes approximately 4-6 months to complete. However, some hospitals and laboratories are now able to generate test results within 3 to 6 weeks. This technology of rapid genetic testing creates new opportunities for providing both women and their treating surgeons with information potentially relevant for deciding between available treatment options, including type of surgery and adjuvant therapy.

The study will focus on newly diagnosed breast cancer patients who, prior to receiving treatment, are identified as having at least a 10% risk of carrying a mutation in the BRCA1 or BRCA2 genes.

We will investigate whether women with a recent diagnosis of breast cancer make use of rapid genetic counseling when offered.

Furthermore, we will investigate whether the process of genetic counseling (and subsequent DNA testing) has influence on the choice of treatment, and whether and how such rapid genetic counseling and testing (RGCT) affects levels of risk perception, cancer-related worries and distress, and decisional satisfaction.

DETAILED DESCRIPTION:
In the Netherlands, approximately 12,000 women are diagnosed with breast cancer annually, of whom about 5-10% carry a mutation in the BRCA1 or BRCA2 gene. Genetic counseling and DNA testing are usually offered to selected patients after primary treatment has been completed (e.g. the first year after diagnosis). For women with a mutation in one of the two breast-ovarian cancer syndrome genes, chances of a second breast cancer are high, and therefore a proportion of these women may opt for preventive measures in addition to their immediate breast cancer treatment. Contralateral prophylactic mastectomy significantly reduces this risk, and is associated with a reduction in mortality. Genetic counseling and testing for breast cancer typically takes approximately 4-6 months to complete.

However, some hospitals and laboratories are now able to generate test results within 3 to 6 weeks. This technology of rapid genetic testing creates new opportunities for providing both women and their treating surgeons with information potentially relevant for deciding between available treatment options, including type of surgery and adjuvant therapy.

The study will focus on newly diagnosed breast cancer patients who, prior to receiving treatment, are identified as having at least a 10% risk of carrying a mutation in the BRCA1 or BRCA2 genes.

We will investigate whether women with a recent diagnosis of breast cancer make use of rapid genetic counseling when offered.

Furthermore, we will investigate whether the process of genetic counseling (and subsequent DNA testing) has influence on the choice of treatment, and whether and how such rapid genetic counseling and testing (RGCT) affects levels of risk perception, cancer-related worries and distress, and decisional satisfaction.

This multicenter study will employ a randomized controlled trial. In an 18 month period newly diagnosed breast cancer patients will be recruited from 13 hospitals in the Amsterdam and Utrecht regions of the Netherlands. Eligible patients will be randomized either to the "usual care" (UC) arm of the study, or to the RGCT arm of the study. The randomization will be done in a ratio of 1:2

Women in the RGCT arm of the study will be referred for genetic counseling within a week after diagnosis, prior to the primary surgery.

Women in the UC condition will receive standard advice and care from their treating physician.

Standardized questionnaires will be administered to all patients at study entry, and at 6 and 12 months to assess all psychosocial outcomes. The endpoints will include:

1. the choice of clinical management strategy, including the uptake of direct bilateral mastectomy (BLM) or of delayed preventive contralateral mastectomy (PCM);
2. cancer risk perception, cancer-related worry and distress;
3. knowledge of genetic aspects of breast cancer;
4. decisional satisfaction; and
5. health-related quality of life (HRQL). The study will also evaluate women's experience of and satisfaction with RGCT (i.e., the timing and quality of the services provided, the perceived impact on treatment decisions, perceived need for additional psychosocial services, etc.). Data on surgical outcomes will be abstracted from the medical records. A subset of women will be interviewed to obtain supplementary, qualitative data about the RGCT experience.

This study will provide essential information about the impact of RGCT on the choice of primary surgical treatment among women with breast cancer with an increased risk that their cancer has a hereditary basis, and about the psychosocial effects of the RGCT process and the ensuing treatment decisions. It will inform clinical geneticists, surgeons and patients about the potential benefits and risks of RGCT, and will be useful in further shaping the content and process of genetic counseling in the diagnostic and early treatment phase of breast cancer.

The study will also yield recommendations for improving the quality of the multidisciplinary care provided in breast cancer clinics by the addition of genetic expertise when patients are at relatively high risk of having a genetic predisposition for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed breast cancer
* 10% or higher chance of carrying BRCA1/2 gene mutation

Exclusion Criteria:

* age <18 years
* does not speak Dutch

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The choice of primary surgical treatment | 1 year

SECONDARY OUTCOMES:
Psychosocial effects | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: N. K. Aaronson, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands

REFERENCES:
- [Derived] Wevers MR, Aaronson NK, Verhoef S, Bleiker EM, Hahn DE, Kuenen MA, van der Sanden-Melis J, Brouwer T, Hogervorst FB, van der Luijt RB, Valdimarsdottir HB, van Dalen T, Theunissen EB, van Ooijen B, de Roos MA, Borgstein PJ, Vrouenraets BC, Vriens E, Bouma WH, Rijna H, Vente JP, Witkamp AJ, Rutgers EJ, Ausems MG. Impact of rapid genetic counselling and testing on the decision to undergo immediate or delayed prophylactic mastectomy in newly diagnosed breast cancer patients: findings from a randomised controlled trial. Br J Cancer. 2014 Feb 18;110(4):1081-7. doi: 10.1038/bjc.2013.805. Epub 2014 Jan 14. PMID 24423928
- [Derived] Wevers MR, Ausems MG, Verhoef S, Bleiker EM, Hahn DE, Hogervorst FB, van der Luijt RB, Valdimarsdottir HB, van Hillegersberg R, Rutgers EJ, Aaronson NK. Behavioral and psychosocial effects of rapid genetic counseling and testing in newly diagnosed breast cancer patients: design of a multicenter randomized clinical trial. BMC Cancer. 2011 Jan 10;11:6. doi: 10.1186/1471-2407-11-6. PMID 21219598